CLINICAL TRIAL: NCT01697462
Title: Evaluation of Safety and Efficacy of Xeloda in Metastatic Colorectal Carcinoma
Brief Title: An Observational Study of Xeloda (Capecitabine) in Patients With Metastatic Colorectal Cancer (AXIOM)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22585
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate the safety and efficacy of Xeloda (capecitabine) administered in monotherapy in patients with metastatic colorectal cancer. Patients will be followed until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Metastatic colorectal cancer
* Receiving Xeloda according to registered indication

Exclusion Criteria:

* Patients who are not eligible for Xeloda treatment according to the Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer
Sampling Method: Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Serbia (4):
  - Belgrade
  - Kamenitz
  - Kragujevac
  - Niš

RESULTS

PARTICIPANT FLOW:
Groups:
- mCRC Participants: Participants who were receiving capecitabine (Xeloda) as per local label for the treatment of metastatic colorectal cancer (mCRC) were followed until progression of the disease (PD), unacceptable toxicity, lost to follow up, death from any cause, or withdrawal of informed consent.
Period: Overall Study
Arm/Group | mCRC Participants
Started | 258
Completed | 181
Not Completed | 77
Not completed — Disease Progression | 1
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 21
Not completed — Withdrawal by Subject | 12
Not completed — Investigator Decision | 21
Not completed — Death | 1
Not completed — Other | 10
Not completed — Missing | 5

BASELINE CHARACTERISTICS:
Population: Baseline population included all enrolled participants.
Groups:
- mCRC Participants: Participants who were receiving capecitabine (Xeloda) as per local label for the treatment of mCRC were followed until PD, unacceptable toxicity, lost to follow up, death from any cause, or withdrawal of informed consent.
Arm/Group | mCRC Participants
Number analyzed (Participants) | 258
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.38 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 151

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-Serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Number of participants with non-serious AEs was exclusive of serious AEs.
Time Frame: Baseline up to end of study (up to 42 months)
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of the study drug and had a subsequent post baseline assessment.
Measure: Number; unit: Participants
Arm/Group | mCRC Participants
Number analyzed (Participants) | 258
Participants
  Non-Serious AEs | 132
  SAEs | 11

2. Secondary Outcome: Percentage of Participants With Disease Progression
Description: Disease progression was defined as greater than 20 percent (%) increase in sum of longest diameter of target lesions compared to baseline.
Time Frame: Baseline to progressive disease or death (up to 42 months)
Population: ITT population. Here, number of participants analyzed (N) signifies those participants who were evaluable for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | mCRC Participants
Number analyzed (Participants) | 257
Percentage of participants | 70.8

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the period from study entry until disease progression or death from any cause. Disease progression was defined as greater than 20% increase in sum of longest diameter of target lesions compared to baseline.
Time Frame: Baseline to progressive disease or death (up to 42 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | mCRC Participants
Number analyzed (Participants) | 257
Months | 4 [3.64 to 4.35]

4. Secondary Outcome: Number of Participants With Hand-Foot Syndrome (HFS)
Description: HFS, also called palmar-plantar erythrodysesthesia, is a side effect or toxicity associated with specific chemotherapy treatments. The National Cancer Institute (2010) describes it as a condition marked by pain, swelling, numbness, tingling, or redness of the hands or feet.
Time Frame: Baseline up to end of study (up to 42 months)
Population: ITT population.
Measure: Number; unit: Participants
Arm/Group | mCRC Participants
Number analyzed (Participants) | 258
Participants | 79

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (up to 42 months)
Arm/Group | mCRC Participants
Serious Adverse Events (participants affected / at risk) | 11/258
Other Adverse Events (participants affected / at risk) | 132/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mCRC Participants (N=258)
Pneumonia (Infections and infestations) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardiotoxicity (Cardiac disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Chest pain (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | mCRC Participants (N=258)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 79
Diarrhoea (Gastrointestinal disorders) | 35
Nausea (Gastrointestinal disorders) | 46
Stomatitis (Gastrointestinal disorders) | 26
Vomiting (Gastrointestinal disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.